CLINICAL TRIAL: NCT04734795
Title: The Prevalence of Dysfunctional Breathing in Children and Adolescents With Asthma
Status: Completed | Type: Observational
Sponsor: Kolding Sygehus (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Signe Vahlkvist, Principal investigator, Kolding Sygehus
Other Study IDs: S-2020-0101-a
Record Dates: First submitted 2021-01-21; First posted 2021-02-02 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Dysfunctional Breathing; Asthma in Children; Asthma
Keywords: Dysfunctional breathing; Asthma in children; Asthma in adolescents
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate the prevalence of dysfunctional breathing in children and adolescents with asthma in a hospital outpatient clinic.

Participants are invited to take the Nijmegen Questionnaire and the Asthma Control Questionnaire. The prevalence of dysfunctional breathing defined as NQ score >= 23 is calculated, and demographics are compared between children with and without dysfunctional breathing.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the prevalence of dysfunctional breathing in children and adolecents with asthma in a hospital outpatient clinic.

Participants are invited to take the Nijmegen Questionnaire and the Asthma Control Questionnaire, during appointments at the outpatient clinic. For this study purpose, each participant only takes the questionnairres once.

Patient data regarding age, sex, asthma medication, lung function, allergic sensitization, method of asthma diagnose, Height, weight and Body mass index is registered from the electronical patient journal.

The prevalence of dysfunctional breathing in the cohort is calculated as the fraction of children with a NQ score >= 23.

The group of children and adolescents with dysfunctional breathing is characterized and compared to the group without dysfunctional breathing, regarding the descriptives mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosed by lung function tests and/or typical symptoms.
* Treatment with inhaled corticosteroids in minimum 3 months.

Exclusion Criteria:

• Other significant cardiopulmonary or muscoluskeletal conditions.

Ages: 10 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children and adolecents with asthma in a hospital outpatient clinic
Sampling Method: Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of children with dysfunctional breathing defined as Nijmegen Questionnaire ( NQ) Score >= 23 | 1 year
  Nijmegen Questionnaire is a 16 point questionnairre addressing dysfunctional breathing. Each question is scored from 0 (best) to 4 (worst). NQ score is summarized between 0-64 points. NQ score >= 23 predicts dysfunctional breathing.

SECONDARY OUTCOMES:
Mask score | 1 year
  Because of the ongoing COVID19 pandemic, face mask is acquired in public, and many children are homeschooled. We therefore generated an 8 question survey about the frequency of wearing mask, breathing difficulties while wearing a mask, and weather there is a lock down of school and sports while survey is taken. Questions are scored from 0-3 points, where 0 is Best and 3 is worst
Asthma Control Questionnaire ( ACQ5) | 1 year
  ACQ5 contains 5 questions regarding asthma symptoms. Each question is scored between 0-6 points, where 0 represents very good asthma control and 6 represents poor asthma control. Total ACQ score is calculates as an average of points.
Age | 1 year
  Age in years of study subjects
Sex | 1 year
  Sex of study subjects
Standardised body mass index (BMI_SDS) | 1 year
  Body mass index is calculated as weight ( kg)/ Height ( m) ^2. As BMI changes with age, BMI standard deviation BMI_SDS is calculated from Danish Reference Material : (Tinggaard J, Aksglaede L, Sørensen K, et al (2014) The 2014 Danish references from birth to 20 years for height, weight and body mass index. Acta Paediatr Int J Paediatr. doi: 10.1111/apa.12468)
The reported use of rescue Beta2 agonist in puffs per week | 1 year
  The reported use of short acting beta 2 agonist in puffs per week the last week.
Forced expiratory volume inthe first second in percent of expected Value. ( FEV1%) | 1 year
  Spirometry is performed according to guidelines. FEV1% is calculated by the spirometry software.
Method of asthma diagnose | 1 year
  Fraction of subjects where asthma was diagnosed objectively from lung function variability (reversibility to beta2 agonist OR positive exercise challenge OR positive mannitol challenge). Method of asthma diagnose is noted from the electronical patient journal

CONTACTS AND LOCATIONS:
Overall Officials: Signe Vahlkvist, Principal Investigator — Kolding Sygehus
Locations (1):
- Kolding Sygehus, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie published results, after deidentification.
Supporting Information: SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to Open@rsyd.dk.
URL: http://open.rsyd.dk